CLINICAL TRIAL: NCT02075840
Title: Randomized, Multicenter, Phase III, Open-Label Study of Alectinib Versus Crizotinib in Treatment-Naive Anaplastic Lymphoma Kinase-Positive Advanced Non-Small Cell Lung Cancer
Brief Title: A Study Comparing Alectinib With Crizotinib in Treatment-Naive Anaplastic Lymphoma Kinase-Positive Advanced Non-Small Cell Lung Cancer Participants
Acronym: ALEX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO28984; 2013-004133-33 (EudraCT Number)
Record Dates: First submitted 2014-02-27; First posted 2014-03-03 (Estimated); Results first posted 2018-03-15 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — alectinib; Crizotinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Alectinib (Experimental): Participants will receive alectinib from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Interventions: Drug: Alectinib
- Crizotinib (Active Comparator): Participants will receive crizotinib from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Interventions: Drug: Crizotinib

INTERVENTIONS:
Drug: Alectinib — Participants will receive alectinib 600 mg orally (four 150 mg capsules) BID from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Other Names: RO5424802
  Arms: Alectinib
Drug: Crizotinib — Participants will receive crizotinib 250 mg capsules orally BID from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
  Arms: Crizotinib

SUMMARY:
This randomized, active controlled, multicenter phase III open-label study is designed to evaluate the efficacy and safety of alectinib compared with crizotinib treatment in participants with treatment-naive anaplastic lymphoma kinase-positive (ALK-positive) advanced non-small cell lung cancer (NSCLC). Participants will be randomized in a 1:1 ratio to receive either alectinib, 600 milligrams (mg) orally twice daily (BID), or crizotinib, 250 mg orally BID. Participants will receive treatment until disease progression, unacceptable toxicity, withdrawal of consent, or death. The study is expected to last approximately 144 months.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed diagnosis of advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC that is ALK-positive as assessed by the Ventana immunohistochemistry (IHC) test
* Life expectancy of at least 12 weeks
* Eastern cooperative oncology group performance status (ECOG PS) of 0-2
* Participants with no prior systemic treatment for advanced or recurrent (Stage IIIB not amenable for multimodality treatment) or metastatic (Stage IV) NSCLC
* Adequate renal, and hematologic function
* Participants must have recovered from effects of any major surgery or significant traumatic injury at least 28 days before the first dose of study treatment
* Measurable disease by response evaluation criteria in solid tumors (RECIST) version 1.1 (v1.1) prior to the administration of study treatment
* Prior brain or leptomeningeal metastases allowed if asymptomatic (e.g., diagnosed incidentally at study baseline)
* Negative pregnancy test for all females of child bearing potential
* Use of highly effective contraception as defined by the study protocol

Exclusion Criteria:

* Participants with a previous malignancy within the past 3 years
* Any gastrointestinal (GI) disorder or liver disease
* National cancer institute common terminology criteria for adverse events (NCI CTCAE) (version 4.0) Grade 3 or higher toxicities due to any prior therapy (e.g., radiotherapy) (excluding alopecia)
* History of organ transplant
* Co-administration of anti-cancer therapies other than those administered in this study
* Participants with baseline QTc greater than (>) 470 milliseconds or symptomatic bradycardia
* Recipient of strong/potent cytochrome P4503A inhibitors or inducers within 14 days prior to the first dose until the end of study treatment
* Recipient of any drug with potential QT interval prolonging effects within 14 days prior to the first dose for all participants and while on treatment through the end of the study for crizotinib-treated participants only
* History of hypersensitivity to any of the additives in the alectinib and crizotinib drug formulation
* Pregnancy or lactation
* Any clinically significant disease or condition (or history of) that could interfere with, or for which the treatment might interfere with, the conduct of the study or the absorption of oral medications or that would, in the opinion of the principal investigator, pose an unacceptable risk to the participant in this study
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol requirements and/or follow-up procedures; those conditions should be discussed with the participant before trial entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 303 (Actual)
Dates: Start 2014-08-19 (Actual); Primary Completion 2017-02-09 (Actual); Study Completion 2025-04-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (98):
- United States (11):
  - North Valley Hem Onc Med Grp, Northridge, California
  - TMPN/ Cancer Care Associates, Redondo Beach, California
  - University of Colorado Cancer Center, Aurora, Colorado
  - University of Miami-Deerfield Beach, Deerfield Beach, Florida
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Med Ctr, Boston, Massachusetts
  - Dana Farber Can Ins, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington Uni School of Medicine, St Louis, Missouri
  - SCRI Oncology Partners, Nashville, Tennessee
  - University of Texas M.D. Anderson Cancer Center, Houston, Texas
- Australia (5):
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Royal North Shore Hospital, St Leonards, New South Wales
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Queen Elizabeth Hospital, Adelaide, South Australia
  - Monash Health Translational Precinct, Victoria, Victoria
- University Clinical Center Sarajevo, Sarajevo, Bosnia and Herzegovina
- Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo, Brazil
- Canada (4):
  - Cross Cancer Institute, Edmonton, Alberta
  - Sunnybrook Odette Cancer Centre, Toronto, Ontario
  - Mount Sinai Hospital, Toronto, Ontario
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Centro Internacional de Estudios Clínicos (CIEC), Santiago, Chile
- China (2):
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Shanghai Pulmonary Hospital, Shanghai
- Clinica CIMCA, San José, Costa Rica
- Kasr Eieny Uni Hospital, Cairo, Egypt
- France (4):
  - Chu Grenoble - Hopital Albert Michallon, Grenoble
  - CHRU de Lille, Lille
  - Centre Leon Berard, Lyon
  - Hopital Haut Leveque, Pessac
- Grupo Angeles, Guatemala City, Guatemala
- Hong Kong (5):
  - Tuen Mun Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Prince of Wales Hosp, Hong Kong
- Israel (2):
  - Rambam Medical Center, Haifa
  - Meir Medical Center, Kfar Saba
- Italy (9):
  - Irccs Ist. Tumori Giovanni Paolo Ii, Bari, Apulia
  - A.O. Universitaria Di Parma, Parma, Emilia-Romagna
  - Ospedale Provinciale Santa Maria Delle Croci, Ravenna, Emilia-Romagna
  - Policlinico Umberto i di Roma, Rome, Lazio
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
  - Azienda Ospedaliero-Universitaria San Luigi Gonzaga, Orbassano, Piedmont
  - Az Ospedaliera Nuovo Garibaldi Quartiere Nesima, Catania, Sicily
  - Azienda Ospedaliera Di Perugia Ospedale s. Maria Della Misericordia, Perugia, Umbria
- Instituto Nacional De Enfermedades Respiratorias, Mexico City, Mexico CITY (federal District), Mexico
- Uni of Auckland, Auckland, New Zealand
- Poland (4):
  - Uniwersyteckie Centrum Kliniczne, Gda?sk
  - Ms Clinsearch Specjalistyczny Niepubliczny Zaklad Opieki Zdrowotnej, Lublin
  - Warminsko-Mazurskie Centrum Chorób P?uc w Olsztynie, Olsztyn
  - Centrum Onkologii - Inst.Im. Marii Sklodowskiej-Curie, Warsaw
- Portugal (3):
  - CHUC - Unidade de Pneumologia Oncológica, Coimbra
  - IPO de Lisboa, Lisbon
  - IPO do Porto, Porto
- Russia (4):
  - Moscow City Oncology Hospital #62, Moscovskaya Oblast, Moscow Oblast
  - SPb City Clin Onc Dsp, Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute named after N.N. Petrov, Saint Petersburg, Sankt-Peterburg
  - N.N.Burdenko Main Military Clinical Hospital, Moscow
- Serbia (2):
  - Clinical Center of Serbia, Belgrade
  - Institute for pulmonary diseases of Vojvodina, Kamenitz
- Singapore (2):
  - National University Hospital, Singapore
  - National Cancer Centre, Singapore
- South Korea (6):
  - National Cancer Center, Gyeonggi-do
  - Seoul National University Bundang Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital General Univ. de Alicante, Alicante
  - Vall d'Hebron Institute of Oncology (VHIO), Barcelona, Barcelona
  - Hospital Universitari Germans Trias i Pujol, Barcelona
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
- Switzerland (4):
  - Universitaetsspital Basel, Basel
  - Inselspital Bern, Bern
  - CHUV, Lausanne
  - UniversitätsSpital Zürich, Zurich
- Taiwan (4):
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung Univ Hosp, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (5):
  - National Cancer Inst., Bangkok
  - Chiang Rai Prachanukroh Hospital, Chiang Rai
  - Khonkaen Hospital, Khonkaen
  - King Chulalongkorn Memorial Hospital, Patumwan
  - Songklanagarind Hospital, Songkhla
- Turkey (Türkiye) (4):
  - Baskent University Adana Dr. Turgut Noyan Practice and Research Hospital, Adana
  - Ankara University Medical Faculty, Ankara
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
- Ukraine (2):
  - Kyiv Regional Oncological Dispensary, Kyiv
  - Lviv State Oncology Regional Treatment and Diagnostic Centre, Lviv
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - University College London Hospital, London
  - Guys & St Thomas Hospital, London

REFERENCES:
- [Derived] Sikkema BJ, Baart SJ, Paats MS, Smit EF, Schols AMWJ, Mathijssen RHJ, van Rossum EFC, Dingemans AC. Body Weight Gain Associated With Alectinib in Patients With ALK+ Non-Small Cell Lung Cancer: Pooled Analysis of Individual Patient Data From Four Prospective Clinical Trials. J Clin Oncol. 2025 Feb 20;43(6):641-650. doi: 10.1200/JCO-24-01579. Epub 2024 Dec 11. PMID 39661917
- [Derived] Dziadziuszko R, Peters S, Mok T, Camidge DR, Gadgeel SM, Ou SI, Konopa K, Noe J, Nowicka M, Bordogna W, Morcos PN, Smoljanovic V, Shaw AT. Circulating Cell-free DNA as a Prognostic Biomarker in Patients with Advanced ALK+ Non-small Cell Lung Cancer in the Global Phase III ALEX Trial. Clin Cancer Res. 2022 May 2;28(9):1800-1808. doi: 10.1158/1078-0432.CCR-21-2840. PMID 35275991
- [Derived] Mok T, Camidge DR, Gadgeel SM, Rosell R, Dziadziuszko R, Kim DW, Perol M, Ou SI, Ahn JS, Shaw AT, Bordogna W, Smoljanovic V, Hilton M, Ruf T, Noe J, Peters S. Updated overall survival and final progression-free survival data for patients with treatment-naive advanced ALK-positive non-small-cell lung cancer in the ALEX study. Ann Oncol. 2020 Aug;31(8):1056-1064. doi: 10.1016/j.annonc.2020.04.478. Epub 2020 May 11. PMID 32418886
- [Derived] Gadgeel S, Peters S, Mok T, Shaw AT, Kim DW, Ou SI, Perol M, Wrona A, Novello S, Rosell R, Zeaiter A, Liu T, Nuesch E, Balas B, Camidge DR. Alectinib versus crizotinib in treatment-naive anaplastic lymphoma kinase-positive (ALK+) non-small-cell lung cancer: CNS efficacy results from the ALEX study. Ann Oncol. 2018 Nov 1;29(11):2214-2222. doi: 10.1093/annonc/mdy405. PMID 30215676
- [Derived] Burudpakdee C, Wong W, Seetasith A, Corvino FA, Yeh W, Gubens M. Economic impact of preventing brain metastases with alectinib in ALK-positive non-small cell lung cancer. Lung Cancer. 2018 May;119:103-111. doi: 10.1016/j.lungcan.2018.03.008. Epub 2018 Mar 9. PMID 29656744
- [Derived] Peters S, Camidge DR, Shaw AT, Gadgeel S, Ahn JS, Kim DW, Ou SI, Perol M, Dziadziuszko R, Rosell R, Zeaiter A, Mitry E, Golding S, Balas B, Noe J, Morcos PN, Mok T; ALEX Trial Investigators. Alectinib versus Crizotinib in Untreated ALK-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Aug 31;377(9):829-838. doi: 10.1056/NEJMoa1704795. Epub 2017 Jun 6. PMID 28586279
- [Derived] Gainor JF, Shaw AT. J-ALEX: alectinib versus crizotinib in ALK-positive lung cancer. Lancet. 2017 Jul 1;390(10089):3-4. doi: 10.1016/S0140-6736(17)31074-7. Epub 2017 May 10. No abstract available. PMID 28501139

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study recruited treatment-naive participants with Anaplastic Lymphoma Kinase (ALK)-positive advanced Non-Small Cell Lung Cancer (NSCLC) in 29 countries from August 2014 to January 2016.
Pre-assignment Details: A total of 303 participants were randomized at the time of clinical cut-off (CCO) date on 9 February 2017 and included in the intent-to-treat (ITT) population; 152 participants in the alectinib arm and 151 participants in the crizotinib arm.
Groups:
- Alectinib: Participants received alectinib at 600 mg orally BID from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
- Crizotinib: Participants received crizotinib at 250 mg orally BID from Visit 0 (baseline) until disease progression, unacceptable toxicity, withdrawal of consent or death.
Period: Overall Study
Arm/Group | Alectinib | Crizotinib
Started | 152 | 151
Completed | 0 | 0
Not Completed | 152 | 151
Not completed — Withdrawal by Subject | 13 | 22
Not completed — Reason not specified | 1 | 0
Not completed — Adverse Event | 0 | 2
Not completed — Death | 35 | 40
Not completed — Lost to Follow-up | 3 | 2
Not completed — Physician Decision | 1 | 3
Not completed — Ongoing at CCOD | 99 | 82

BASELINE CHARACTERISTICS:
Population: Analysis was performed on intent to treat (ITT) population which included all randomized participants in the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Alectinib | Crizotinib | Total
Number analyzed (Participants) | 152 | 151 | 303
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.3 (12.0) | 53.8 (13.5) | 55.1 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 87 | 171
  Male | 68 | 64 | 132
Race/Ethnicity, Customized [Number; unit: Participants]
  Ethnicity - Hispanic or Latino | 8 | 8 | 16
  Ethinicity - Not Hispanic or Latino | 138 | 136 | 274
  Ethnicity - Not Stated | 6 | 7 | 13
Race/Ethnicity, Customized [Number; unit: Participants]
  Race - American Indian or Alaska Native | 4 | 0 | 4
  Race - Asian | 69 | 69 | 138
  Race - Black or African American | 0 | 4 | 4
  Race - Native Hawaiian or other Pacific Islander | 1 | 1 | 2
  Race - White | 76 | 75 | 151
  Race - Unknown | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) by Investigator Assessment
Description: PFS was assessed as time to disease progression or death whichever occurred first by investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) Criteria. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 millimeter (mm) and the appearance of new lesions.
Time Frame: Randomization to first documented disease progression or death, whichever occurs first (assessed every 8 weeks up to 33 months)
Population: ITT population included all randomized participants in the study. Number of participants analyzed is the total participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
months | NA [17.7 to NA] — The median PFS had not been reached in the alectinib arm at the time of data cutoff date (9 Feb 2017). | 11.1 [9.1 to 13.1]
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Stratified hazard ratio and p-value are stratified for covariates Race (Asian vs Non-Asian) and CNS metastases at baseline by IRC; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio, stratified = 0.47, 95% CI 2-sided [0.34 to 0.65]

2. Primary Outcome: Percentage of Participants With PFS Event by Investigator Assessment
Description: PFS was assessed percentage of participants with disease progression or death whichever occurred first by investigator assessment using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) Criteria. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 millimeter (mm) and the appearance of new lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 40.8 | 67.5

3. Secondary Outcome: PFS Independent Review Committee (IRC)-Assessed
Description: PFS was assessed as time to disease progression or death whichever occurred first by IRC assessment using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) Criteria. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm and the appearance of new lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
months | 25.7 [19.9 to NA] — The upper limit of the CI could not be estimated in the alectinib arm at the time of data cutoff date (9 Feb 2017). | 10.4 [7.7 to 14.6]
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Test type: Superiority; p < 0.0001, Log Rank; Stratified hazard ratio and p-value are stratified for covariates Race (Asian vs Non-Asian) and CNS metastases at baseline by IRC; Hazard Ratio (HR) = 0.50, 95% CI 2-sided [0.36 to 0.70]

4. Secondary Outcome: Percentage of Participants With PFS Event by IRC
Description: PFS was assessed as percentage of participants with disease progression or death whichever occurred first by IRC assessment using Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 (v1.1) Criteria. As per RECIST v1.1, disease progression is a 20% increase in the sum of the diameters of target lesions, an increase in size of measurable lesions by at least 5 mm and the appearance of new lesions.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 41.4 | 60.9

5. Secondary Outcome: Percentage of Participants With Central Nervous System (CNS) Progression as Determined by IRC Using RECIST V1.1 Criteria
Description: CNS progression was assessed as percentage of participants with an event defined as time from randomization until first radiographic evidence of CNS progression by IRC. The risk for a CNS progression without a prior non-CNS progression with alectinib compared with crizotinib.
Time Frame: Randomization to CNS PD as first occurrence of disease progression (assessed every 8 weeks up to 33 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 11.8 | 45.0
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Test type: Superiority — IRC, RECIST v1.1 Stratified Analysis (by race (Asian vs non-Asian) and CNS metastases at baseline by IRC); p < 0.0001, Log Rank; Cause-Specific Hazard Ratio = 0.16, 95% CI 2-sided [0.10 to 0.28]

6. Secondary Outcome: Percentage of Participants With Central Nervous System (CNS) Progression as Determined by IRC Using Revised Assessment in Neuro Oncology (RANO) Criteria
Description: CNS progression was assessed as percentage of participants with event defined as time from randomization until first radiographic evidence of CNS progression by IRC. The risk for a CNS progression without a prior non-CNS progression with alectinib compared with crizotinib.
Time Frame: Randomization to the first occurrence of disease progression in the CNS (assessed every 8 weeks up to 33 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 10.5 | 35.8

7. Secondary Outcome: Percentage of Participants With Objective Response Rate (ORR) of Complete Response (CR) or Partial Response (PR) as Determined by The Investigators According to RECIST V1.1 Criteria
Description: ORR was defined as the percentage of participants who attained CR or PR. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 82.9 [75.95 to 88.51] | 75.5 [67.84 to 82.12]
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Test type: Superiority; p = 0.0936, Mantel Haenszel — Stratified analysis; Difference in Overall Response Rates = 7.40, 95% CI 2-sided [-1.71 to 16.50]

8. Secondary Outcome: Duration of Response (DOR) According to RECIST V1.1 Criteria as Assessed by the Investigators
Description: DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death, whichever occurred first. DOR was evaluated for participants who had a best overall response (BOR) of CR or PR.
Time Frame: First occurrence of objective response to first documented disease progression or death, whichever occurs first (assessed every 8 weeks up to 33 months)
Population: ITT population included all participants randomized in the study, irrespective of whether or not they received study drug. Number analyzed indicates number of participants with a BOR of CR or PR.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Months | NA [NA to NA] — The median DOR was not estimable [95% CI: NE] in the alectinib arm due to the low number of contributing events of disease progression or death. | 11.1 [7.9 to 13.0]

9. Secondary Outcome: Overall Survival (OS)
Description: Overall survival (OS) was defined as the time from randomization to death from any cause.
Time Frame: From randomization until death (up to 43 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
months | NA [NA to NA] — Median time to OS event was not reached in participants in either treatment arm at the time of data cutoff (9 Feb 2017). | NA [NA to NA] — Median time to OS event was not reached in participants in either treatment arm at the time of data cutoff (9 Feb 2017).
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Test type: Superiority; p = 0.2405, Log Rank — Stratified analysis; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.48 to 1.20]

10. Secondary Outcome: Percentage of Participants With OS Event
Description: Overall survival (OS) was defined as the time from randomization to death from any cause.
Time Frame: From randomization until death (up to 43 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 23.0 | 26.5

11. Secondary Outcome: Percentage of Participants With CNS ORR of CR or PR IRC-assessed According to RECIST v1.1 Criteria
Description: CNS ORR was defined as the percentage of participants who attained CR or PR and had measurable/non-measurable CNS lesions at baseline. As per RECIST v1.1, CR: Disappearance of all target lesions and any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm, PR: At least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum of diameters.
Time Frame: as for outcome 1
Population: ITT population included all randomized participants in the study. Number of participants analyzed is the total participants who were evaluable for this outcome measure (number of participants with measurable/non-measurable CNS lesions at baseline).
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants
  Measurable CNS lesions at baseline: number analyzed (Participants) | 21 | 22
  Measurable CNS lesions at baseline | 81.0 [58.09 to 94.55] | 50.0 [28.22 to 71.78]
  Measurable and non-measurable CNS lesions: number analyzed (Participants) | 64 | 58
  Measurable and non-measurable CNS lesions | 59.4 [46.37 to 71.49] | 25.9 [15.26 to 39.04]

12. Secondary Outcome: CNS DOR IRC-assessed According to RECIST v1.1 Criteria
Description: CNS DOR was defined as the time from when response (CR or PR) was first documented to first documented disease progression or death, whichever occurred first. DOR was evaluated for participants who had a best overall response (BOR) of CR or PR.
Time Frame: First occurrence of CNS objective response to first documented disease progression or death, whichever occurs first (assessed every 8 weeks up to 33 months)
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 21 | 22
months | 17.3 [14.8 to NA] — The upper limit of the CI for CNS DOR could not be estimated at time of the data cutoff for participants in the alectinib arm. | 5.5 [2.1 to 17.3]

13. Secondary Outcome: Percentage of Participants With Adverse Events
Description: An adverse event (AE) is any untoward medical occurrence in a participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.
Time Frame: Baseline up to 28 months in the crizotinib arm and up to 30 months in the alectinib arm
Population: Safety (SAF) population included all participants who received at least one dose of any study drug.
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants | 97.0 | 97.0

14. Secondary Outcome: Area Under The Concentration-Time Curve (AUC) of Alectinib
Time Frame: Pre-dose (within 2 hours before alectinib) (baseline), 1, 2, 4, 6, and 8 hours post-dose at Visit 0 (first dosing day) and Week 4; Pre-dose (within 2 hours) at Week 8, then every 8 weeks until disease progression or death/withdrawal (up to 33 months)
Population: The Pharmacokinetic (PK) Evaluable Population included all participants who received any dose of alectinib and who had at least one post-baseline PK sample available.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 144
hr*ng/mL
  Baseline: number analyzed (Participants) | 10
  Baseline | 713 (104.9)
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 5030 (47.2)

15. Secondary Outcome: Maximum Concentration (Cmax) of Alectinib
Time Frame: Pre-dose (within 2 hours before alectinib), 1, 2, 4, 6, and 8 hours post-dose at baseline and Week 4; Pre-dose (within 2 hours before alectinib) at Week 8, then every 8 weeks until disease progression or death/withdrawal from study (up to 33 months)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Alectinib
Number analyzed (Participants) | 144
nanogram/milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 10
  Baseline | 211 (55.5)
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 717 (46.8)

16. Secondary Outcome: Time to Reach Cmax (Tmax) of Alectinib
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Alectinib
Number analyzed (Participants) | 144
hours
  Baseline: number analyzed (Participants) | 10
  Baseline | 6.03 [1.98 to 12.00]
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 4.02 [2.00 to 8.00]

17. Secondary Outcome: AUC of Alectinib Metabolite
Time Frame: as for outcome 14
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hr*ng/mL
Arm/Group | Alectinib
Number analyzed (Participants) | 144
hr*ng/mL
  Baseline: number analyzed (Participants) | 10
  Baseline | 142 (191.7)
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 2230 (37.0)

18. Secondary Outcome: Cmax of Alectinib Metabolite
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram/milliliter (ng/mL)
Arm/Group | Alectinib
Number analyzed (Participants) | 144
nanogram/milliliter (ng/mL)
  Baseline: number analyzed (Participants) | 10
  Baseline | 56.2 (80.1)
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 321 (32.0)

19. Secondary Outcome: Tmax of Alectinib Metabolite
Time Frame: as for outcome 15
Population: as for outcome 14
Measure: Median (Full Range); unit: hours
Arm/Group | Alectinib
Number analyzed (Participants) | 144
hours
  Baseline: number analyzed (Participants) | 10
  Baseline | 8.00 [5.98 to 12.00]
  Treatment - week 4: number analyzed (Participants) | 9
  Treatment - week 4 | 6.00 [2.00 to 10.00]

20. Secondary Outcome: Time to Deterioration by European Organization for The Research And Treatment of Cancer (EORTC) Quality Of Life Questionnaire Core 30 (C30)
Description: The EORTC QLQ-30 module generated one multiple-item scale score assessing dyspnea and a series of single item scores assessing chest pain, arm/shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning. Confirmed clinically meaningful deterioration in global health status or function is defined as a >or=10-point decrease from baseline in a symptom score that must be held for at least two consecutive assessments or an initial >or=10-point decrease from baseline followed by death within 5 weeks from the last assessment.
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
months
  Fatigue | NA [NA to NA] — Median deterioration not reached at CCOD | NA [9.4 to NA] — Median deterioration not reached at CCOD
  Dyspnea | NA [NA to NA] — Median deterioration not reached at CCOD | NA [NA to NA] — Median deterioration not reached at CCOD
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Fatigue; Test type: Superiority; p = 0.2079, Log Rank; Stratified analysis; Hazard Ratio (HR) = 0.74, 95% CI 2-sided [0.46 to 1.19]
Statistical Analysis 2: Comparison: Alectinib vs Crizotinib; Dyspnea; Test type: Superiority; p = 0.1137, Log Rank — Stratified analysis; Hazard Ratio (HR) = 1.66, 95% CI 2-sided [0.88 to 3.15]

21. Secondary Outcome: Percentage of Participants With Deterioration by EORTC Quality Of Life Questionnaire Core 30 (C30)
Description: as for outcome 20
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants
  Fatigue | 21.7 | 25.2
  Dyspnea | 17.1 | 9.9

22. Secondary Outcome: Time to Deterioration by EORTC Quality of Life Questionnaire Lung Cancer Module 13 (LC13)
Description: The EORTC QLQ-LC13 module generated one multiple-item scale score assessing dyspnea and a series of single item scores assessing chest pain, arm/shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning. Confirmed clinically meaningful deterioration in lung cancer symptoms is defined as a >or=10-point increase from baseline in a symptom score that must be held for at least two consecutive assessments or an initial >or=10-point increase above baseline followed by death within 5 weeks from the last assessment.
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
months
  Coughing | NA [24.0 to NA] — Median deterioration not reached at CCOD | NA [NA to NA] — Median deterioration not reached at CCOD
  Dyspnea | 22.8 [11.8 to NA] — Upper limit of the CI not reached at CCOD | NA [21.0 to NA] — Median deterioration not reached at CCOD
  Pain in arm and shoulder | NA [NA to NA] — Median deterioration not reached at CCOD | NA [NA to NA] — Median deterioration not reached at CCOD
  Pain in chest | NA [NA to NA] — Median deterioration not reached at CCOD | NA [NA to NA] — Median deterioration not reached at CCOD
  Composite score (c, p in c, d) | 12.7 [5.0 to NA] — Upper limit of the CI not reached at CCOD | 21.0 [9.8 to NA] — Upper limit of the CI not reached at CCOD
Statistical Analysis 1: Comparison: Alectinib vs Crizotinib; Coughing; Test type: Superiority; p = 0.7042, Log Rank — Stratified analysis; Hazard Ratio (HR) = 0.88, 95% CI 2-sided [0.44 to 1.74]
Statistical Analysis 2: Comparison: Alectinib vs Crizotinib; Dyspnea; Test type: Superiority; p = 0.0285, Log Rank — Stratified analysis; Hazard Ratio (HR) = 1.76, 95% CI 2-sided [1.05 to 2.92]
Statistical Analysis 3: Comparison: Alectinib vs Crizotinib; Pain in arm and shoulder; Test type: Superiority; p = 0.2377, Log Rank — Stratified analysis; Hazard Ratio (HR) = 1.43, 95% CI 2-sided [0.79 to 2.61]
Statistical Analysis 4: Comparison: Alectinib vs Crizotinib; Pain in chest; Test type: Superiority; p = 0.0796, Log Rank — Stratified analysis; Hazard Ratio (HR) = 0.51, 95% CI 2-sided [0.24 to 1.10]
Statistical Analysis 5: Comparison: Alectinib vs Crizotinib; Composite score; Test type: Superiority; p = 0.6435, Log Rank — Stratified analysis; Hazard Ratio (HR) = 1.10, 95% CI 2-sided [0.72 to 1.68]

23. Secondary Outcome: Percentage of Participants With Deterioration by EORTC Quality of Life Questionnaire Lung Cancer Module 13 (LC13)
Description: as for outcome 22
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Percentage of Participants
  Coughing | 11 | 11
  Dyspnea | 28 | 16
  Pain in arm and shoulder | 18 | 12
  Pain in chest | 7 | 11
  Composite score (c, p in c, d) | 32 | 28

24. Secondary Outcome: Health-Related Quality of Life (HRQoL) by EORTC Quality of Life Questionnaire C30 Score
Description: The EORTC QLQ-C30 questionnaire consisted of 30 questions generating five functional scores (physical, role, cognitive, emotional, and social); a global health status/global quality of life scale score; three symptom scale scores (fatigue, pain, and nausea and vomiting); and six stand alone one-item scores that capture additional symptoms (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea) and perceived financial burden. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning.
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: ITT population included all participants randomized in the study, irrespective of whether or not they received study drug. Number analyzed indicates number of participants evaluated for specified time points.
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Score on a scale
  Baseline: number analyzed (Participants) | 100 | 97
  Baseline | 66.67 [8.3 to 100.0] | 66.67 [0.0 to 100.0]
  Treatment - week 4: number analyzed (Participants) | 95 | 89
  Treatment - week 4 | 66.67 [0.0 to 100.0] | 66.67 [16.7 to 100.0]
  Treatment - week 8: number analyzed (Participants) | 89 | 84
  Treatment - week 8 | 75.0 [16.7 to 100.0] | 75.0 [16.7 to 100.0]
  Treatment - week 12: number analyzed (Participants) | 75 | 78
  Treatment - week 12 | 75.0 [25.0 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 16: number analyzed (Participants) | 79 | 73
  Treatment - week 16 | 75.0 [16.7 to 100.0] | 83.33 [16.7 to 100.0]
  Treatment - week 20: number analyzed (Participants) | 73 | 67
  Treatment - week 20 | 75.0 [16.7 to 100.0] | 75.0 [16.7 to 100.0]
  Treatment - week 24: number analyzed (Participants) | 77 | 71
  Treatment - week 24 | 75.0 [16.7 to 100.0] | 83.33 [8.3 to 100.0]
  Treatment - week 28: number analyzed (Participants) | 67 | 62
  Treatment - week 28 | 75.0 [33.3 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 32: number analyzed (Participants) | 73 | 65
  Treatment - week 32 | 75.0 [33.3 to 100.0] | 66.67 [8.3 to 100.0]
  Treatment - week 36: number analyzed (Participants) | 64 | 61
  Treatment - week 36 | 79.17 [16.7 to 100.0] | 66.67 [16.7 to 100.0]
  Treatment - week 40: number analyzed (Participants) | 74 | 50
  Treatment - week 40 | 75.0 [16.7 to 100.0] | 83.33 [33.3 to 100.0]
  Treatment - week 44: number analyzed (Participants) | 62 | 47
  Treatment - week 44 | 83.33 [16.7 to 100.0] | 83.33 [16.7 to 100.0]
  Treatment - week 48: number analyzed (Participants) | 67 | 47
  Treatment - week 48 | 66.67 [25.0 to 100.0] | 83.33 [41.7 to 100.0]
  Treatment - week 52: number analyzed (Participants) | 58 | 44
  Treatment - week 52 | 83.33 [16.7 to 100.0] | 75.00 [41.7 to 100.0]
  Treatment - week 56: number analyzed (Participants) | 61 | 48
  Treatment - week 56 | 75.0 [16.7 to 100.0] | 75.0 [41.7 to 100.0]
  Treatment - week 60: number analyzed (Participants) | 47 | 39
  Treatment - week 60 | 75.0 [33.3 to 100.0] | 75.0 [50.0 to 100.0]
  Treatment - week 64: number analyzed (Participants) | 55 | 39
  Treatment - week 64 | 75.0 [33.3 to 100.0] | 83.33 [41.7 to 100.0]
  Treatment - week 68: number analyzed (Participants) | 49 | 34
  Treatment - week 68 | 75.0 [33.3 to 100.0] | 79.17 [33.3 to 100.0]
  Treatment - week 72: number analyzed (Participants) | 54 | 34
  Treatment - week 72 | 75.0 [33.3 to 100.0] | 75.00 [8.3 to 100.0]
  Treatment - week 76: number analyzed (Participants) | 42 | 29
  Treatment - week 76 | 75.0 [41.7 to 100.0] | 75.0 [16.7 to 100.0]
  Treatment - week 80: number analyzed (Participants) | 43 | 23
  Treatment - week 80 | 75.0 [33.3 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 84: number analyzed (Participants) | 33 | 19
  Treatment - week 84 | 83.33 [41.7 to 100.0] | 66.67 [33.3 to 100.0]
  Treatment - week 88: number analyzed (Participants) | 36 | 16
  Treatment - week 88 | 75.0 [33.3 to 100.0] | 66.67 [33.3 to 100.0]
  Treatment - week 92: number analyzed (Participants) | 30 | 13
  Treatment - week 92 | 70.83 [33.3 to 100.0] | 75.0 [50.0 to 100.0]
  Treatment - week 96: number analyzed (Participants) | 22 | 11
  Treatment - week 96 | 66.67 [33.3 to 100.0] | 66.67 [33.3 to 100.0]
  Treatment - week 100: number analyzed (Participants) | 18 | 10
  Treatment - week 100 | 66.67 [25.0 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 104: number analyzed (Participants) | 15 | 7
  Treatment - week 104 | 66.67 [50.0 to 100.0] | 66.67 [50.0 to 100.0]
  Treatment - week 108: number analyzed (Participants) | 11 | 7
  Treatment - week 108 | 66.67 [50.0 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 112: number analyzed (Participants) | 9 | 4
  Treatment - week 112 | 75.0 [50.0 to 100.0] | 75.0 [33.3 to 100.0]
  Treatment - week 116: number analyzed (Participants) | 4 | 2
  Treatment - week 116 | 70.83 [41.7 to 100.0] | 91.67 [83.3 to 100.0]
  Treatment - week 120: number analyzed (Participants) | 3 | 151
  Treatment - week 120 | 83.3 [50.0 to 100.0] | NA [NA to NA] — Not evaluable at week 120

25. Secondary Outcome: HRQoL by EORTC Quality of Life Questionnaire LC13 Score Coughing
Description: The EORTC QLQ-LC13 module generated one multiple-item scale score assessing dyspnea and a series of single item scores assessing chest pain, arm/shoulder pain, pain in other parts, coughing, sore mouth, dysphagia, peripheral neuropathy, alopecia, and hemoptysis. All the scales and single-item scores were linearly transformed so that each score ranged from 0 to 100. A higher score on the global health and functioning subscales is indicative of better functioning.
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 24
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Score on a scale
  Baseline: number analyzed (Participants) | 100 | 96
  Baseline | 33.33 [0.0 to 100.0] | 33.33 [0.0 to 100.0]
  Treatment - week 4: number analyzed (Participants) | 95 | 89
  Treatment - week 4 | 33.33 [0.0 to 100.0] | 33.33 [0.0 to 100.0]
  Treatment - week 8: number analyzed (Participants) | 89 | 84
  Treatment - week 8 | 33.33 [0.0 to 66.7] | 33.33 [0.0 to 100.0]
  Treatment - week 12: number analyzed (Participants) | 75 | 78
  Treatment - week 12 | 33.33 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - week 16: number analyzed (Participants) | 79 | 73
  Treatment - week 16 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - week 20: number analyzed (Participants) | 73 | 67
  Treatment - week 20 | 33.33 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - week 24: number analyzed (Participants) | 77 | 71
  Treatment - week 24 | 33.33 [0.0 to 100.0] | 33.33 [0.0 to 100.0]
  Treatment - week 28: number analyzed (Participants) | 67 | 62
  Treatment - week 28 | 33.33 [0.0 to 100.0] | 16.67 [0.0 to 100.0]
  Treatment - week 32: number analyzed (Participants) | 73 | 65
  Treatment - week 32 | 33.33 [0.0 to 100.0] | 33.33 [0.0 to 100.0]
  Treatment - week 36: number analyzed (Participants) | 64 | 61
  Treatment - week 36 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - week 40: number analyzed (Participants) | 74 | 50
  Treatment - week 40 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 44: number analyzed (Participants) | 62 | 47
  Treatment - week 44 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 48: number analyzed (Participants) | 67 | 47
  Treatment - week 48 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 52: number analyzed (Participants) | 58 | 44
  Treatment - week 52 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - week 56: number analyzed (Participants) | 61 | 48
  Treatment - week 56 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - week 60: number analyzed (Participants) | 47 | 39
  Treatment - week 60 | 33.33 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - week 64: number analyzed (Participants) | 55 | 39
  Treatment - week 64 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 68: number analyzed (Participants) | 49 | 34
  Treatment - week 68 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 72: number analyzed (Participants) | 54 | 34
  Treatment - week 72 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 76: number analyzed (Participants) | 42 | 29
  Treatment - week 76 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 80: number analyzed (Participants) | 43 | 23
  Treatment - week 80 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 33.33]
  Treatment - week 84: number analyzed (Participants) | 33 | 19
  Treatment - week 84 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.33]
  Treatment - week 88: number analyzed (Participants) | 36 | 16
  Treatment - week 88 | 33.33 [0.0 to 100.0] | 0.0 [0.0 to 33.33]
  Treatment - week 92: number analyzed (Participants) | 30 | 13
  Treatment - week 92 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - week 96: number analyzed (Participants) | 22 | 11
  Treatment - week 96 | 16.67 [0.0 to 66.7] | 0.0 [0.0 to 33.33]
  Treatment - week 100: number analyzed (Participants) | 18 | 10
  Treatment - week 100 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 33.3]
  Treatment - week 104: number analyzed (Participants) | 15 | 7
  Treatment - week 104 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - week 108: number analyzed (Participants) | 11 | 7
  Treatment - week 108 | 33.33 [0.0 to 66.7] | 33.33 [0.0 to 33.33]
  Treatment - week 112: number analyzed (Participants) | 9 | 4
  Treatment - week 112 | 33.33 [0.0 to 33.33] | 0.0 [0.0 to 33.33]
  Treatment - week 116: number analyzed (Participants) | 4 | 2
  Treatment - week 116 | 33.33 [0.0 to 33.33] | 16.67 [0.0 to 33.33]
  Treatment - week 120: number analyzed (Participants) | 3 | 0
  Treatment - week 120 | 33.33 [33.33 to 33.33] |

26. Secondary Outcome: HRQoL by EORTC Quality of Life Questionnaire LC13 Score Dyspnoea
Description: as for outcome 25
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 24
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Score on a scale
  Baseline: number analyzed (Participants) | 100 | 96
  Baseline | 22.22 [0.0 to 100.0] | 22.22 [0.0 to 100.0]
  Treatment - Week 4: number analyzed (Participants) | 95 | 89
  Treatment - Week 4 | 22.22 [0.0 to 100.0] | 22.22 [0.0 to 88.9]
  Treatment - Week 8: number analyzed (Participants) | 89 | 84
  Treatment - Week 8 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 66.7]
  Treatment - Week 12: number analyzed (Participants) | 75 | 78
  Treatment - Week 12 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 66.7]
  Treatment - Week 16: number analyzed (Participants) | 79 | 73
  Treatment - Week 16 | 22.22 [0.0 to 77.8] | 11.11 [0.0 to 88.9]
  Treatment - Week 20: number analyzed (Participants) | 73 | 67
  Treatment - Week 20 | 22.22 [0.0 to 88.9] | 11.11 [0.0 to 66.7]
  Treatment - Week 24: number analyzed (Participants) | 77 | 71
  Treatment - Week 24 | 22.22 [0.0 to 77.8] | 11.11 [0.0 to 77.8]
  Treatment - Week 28: number analyzed (Participants) | 67 | 62
  Treatment - Week 28 | 11.11 [0.0 to 44.4] | 11.11 [0.0 to 100.0]
  Treatment - Week 32: number analyzed (Participants) | 73 | 65
  Treatment - Week 32 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 88.9]
  Treatment - Week 36: number analyzed (Participants) | 64 | 61
  Treatment - Week 36 | 16.67 [0.0 to 77.8] | 11.11 [0.0 to 66.7]
  Treatment - Week 40: number analyzed (Participants) | 74 | 50
  Treatment - Week 40 | 11.11 [0.0 to 55.6] | 5.56 [0.0 to 66.7]
  Treatment - Week 44: number analyzed (Participants) | 62 | 47
  Treatment - Week 44 | 11.11 [0.0 to 88.9] | 11.11 [0.0 to 77.8]
  Treatment - Week 48: number analyzed (Participants) | 67 | 47
  Treatment - Week 48 | 22.22 [0.0 to 55.6] | 11.11 [0.0 to 44.4]
  Treatment - Week 52: number analyzed (Participants) | 58 | 44
  Treatment - Week 52 | 22.22 [0.0 to 44.4] | 11.11 [0.0 to 66.7]
  Treatment - Week 56: number analyzed (Participants) | 61 | 48
  Treatment - Week 56 | 22.22 [0.0 to 77.8] | 11.11 [0.0 to 77.8]
  Treatment - Week 60: number analyzed (Participants) | 47 | 39
  Treatment - Week 60 | 22.22 [0.0 to 77.8] | 0.0 [0.0 to 55.6]
  Treatment - Week 64: number analyzed (Participants) | 55 | 39
  Treatment - Week 64 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 66.7]
  Treatment - Week 68: number analyzed (Participants) | 49 | 34
  Treatment - Week 68 | 22.22 [0.0 to 77.8] | 11.11 [0.0 to 55.6]
  Treatment - Week 72: number analyzed (Participants) | 54 | 34
  Treatment - Week 72 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 44.4]
  Treatment - Week 76: number analyzed (Participants) | 42 | 29
  Treatment - Week 76 | 11.11 [0.0 to 66.7] | 11.11 [0.0 to 55.6]
  Treatment - Week 80: number analyzed (Participants) | 43 | 23
  Treatment - Week 80 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 55.6]
  Treatment - Week 84: number analyzed (Participants) | 33 | 19
  Treatment - Week 84 | 11.11 [0.0 to 66.7] | 11.11 [0.0 to 44.4]
  Treatment - Week 88: number analyzed (Participants) | 36 | 16
  Treatment - Week 88 | 22.22 [0.0 to 55.6] | 22.22 [0.0 to 33.3]
  Treatment - Week 92: number analyzed (Participants) | 30 | 13
  Treatment - Week 92 | 22.22 [0.0 to 44.4] | 22.22 [0.0 to 77.8]
  Treatment - Week 96: number analyzed (Participants) | 22 | 11
  Treatment - Week 96 | 22.22 [0.0 to 66.7] | 22.22 [0.0 to 44.4]
  Treatment - Week 100: number analyzed (Participants) | 18 | 10
  Treatment - Week 100 | 22.22 [0.0 to 55.6] | 27.78 [0.0 to 44.4]
  Treatment - Week 104: number analyzed (Participants) | 15 | 7
  Treatment - Week 104 | 11.11 [0.0 to 66.7] | 11.11 [0.0 to 33.3]
  Treatment - Week 108: number analyzed (Participants) | 11 | 7
  Treatment - Week 108 | 22.22 [0.0 to 66.7] | 11.11 [0.0 to 33.3]
  Treatment - Week 112: number analyzed (Participants) | 9 | 4
  Treatment - Week 112 | 11.11 [11.11 to 44.4] | 27.78 [0.0 to 33.3]
  Treatment - Week 116: number analyzed (Participants) | 4 | 2
  Treatment - Week 116 | 16.67 [11.1 to 22.2] | 16.67 [0.0 to 33.3]
  Treatment - Week 120: number analyzed (Participants) | 3 | 0
  Treatment - Week 120 | 22.22 [11.1 to 33.3] |

27. Secondary Outcome: HRQoL by EORTC Quality of Life Questionnaire LC13 Score Pain in Chest
Description: as for outcome 25
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 24
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Score on a scale
  Baseline: number analyzed (Participants) | 100 | 96
  Baseline | 33.33 [0.0 to 100.0] | 0.0 [0.0 to 100.0]
  Treatment - Week 4: number analyzed (Participants) | 95 | 89
  Treatment - Week 4 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 8: number analyzed (Participants) | 89 | 84
  Treatment - Week 8 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 66.7]
  Treatment - Week 12: number analyzed (Participants) | 75 | 78
  Treatment - Week 12 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 16: number analyzed (Participants) | 79 | 73
  Treatment - Week 16 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 66.7]
  Treatment - Week 20: number analyzed (Participants) | 73 | 67
  Treatment - Week 20 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 24: number analyzed (Participants) | 77 | 71
  Treatment - Week 24 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 66.7]
  Treatment - Week 28: number analyzed (Participants) | 67 | 62
  Treatment - Week 28 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 32: number analyzed (Participants) | 73 | 65
  Treatment - Week 32 | 0.00 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 36: number analyzed (Participants) | 64 | 61
  Treatment - Week 36 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 40: number analyzed (Participants) | 74 | 50
  Treatment - Week 40 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 44: number analyzed (Participants) | 62 | 47
  Treatment - Week 44 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - Week 48: number analyzed (Participants) | 67 | 47
  Treatment - Week 48 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 52: number analyzed (Participants) | 58 | 44
  Treatment - Week 52 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 56: number analyzed (Participants) | 61 | 48
  Treatment - Week 56 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 60: number analyzed (Participants) | 47 | 39
  Treatment - Week 60 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 66.7]
  Treatment - Week 64: number analyzed (Participants) | 55 | 39
  Treatment - Week 64 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 68: number analyzed (Participants) | 49 | 34
  Treatment - Week 68 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 72: number analyzed (Participants) | 54 | 34
  Treatment - Week 72 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 76: number analyzed (Participants) | 42 | 29
  Treatment - Week 76 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 80: number analyzed (Participants) | 43 | 23
  Treatment - Week 80 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 84: number analyzed (Participants) | 33 | 19
  Treatment - Week 84 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 88: number analyzed (Participants) | 36 | 16
  Treatment - Week 88 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 92: number analyzed (Participants) | 30 | 13
  Treatment - Week 92 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 33.3]
  Treatment - Week 96: number analyzed (Participants) | 22 | 11
  Treatment - Week 96 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 100: number analyzed (Participants) | 18 | 10
  Treatment - Week 100 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 104: number analyzed (Participants) | 15 | 7
  Treatment - Week 104 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 108: number analyzed (Participants) | 11 | 7
  Treatment - Week 108 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 112: number analyzed (Participants) | 9 | 4
  Treatment - Week 112 | 0.0 [0.0 to 66.7] | 16.67 [0.0 to 33.3]
  Treatment - Week 116: number analyzed (Participants) | 4 | 2
  Treatment - Week 116 | 0.0 [0.0 to 33.3] | 16.67 [0.0 to 33.3]
  Treatment - Week 120: number analyzed (Participants) | 3 | 0
  Treatment - Week 120 | 0.0 [0.0 to 66.7] |

28. Secondary Outcome: HRQoL by EORTC Quality of Life Questionnaire LC13 Score Pain in Arm and Shoulder
Description: as for outcome 25
Time Frame: Baseline, every 4 weeks until disease progression (up to 33 months)
Population: as for outcome 24
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Alectinib | Crizotinib
Number analyzed (Participants) | 152 | 151
Score on a scale
  Baseline: number analyzed (Participants) | 100 | 96
  Baseline | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 100.0]
  Treatment - Week 4: number analyzed (Participants) | 95 | 89
  Treatment - Week 4 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - Week 8: number analyzed (Participants) | 89 | 84
  Treatment - Week 8 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - Week 12: number analyzed (Participants) | 75 | 78
  Treatment - Week 12 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - Week 16: number analyzed (Participants) | 79 | 73
  Treatment - Week 16 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 20: number analyzed (Participants) | 73 | 67
  Treatment - Week 20 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 24: number analyzed (Participants) | 77 | 71
  Treatment - Week 24 | 0.0 [0.0 to 33.3] | 0.0 [0.0 to 66.7]
  Treatment - Week 28: number analyzed (Participants) | 67 | 62
  Treatment - Week 28 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 32: number analyzed (Participants) | 73 | 65
  Treatment - Week 32 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - Week 36: number analyzed (Participants) | 64 | 61
  Treatment - Week 36 | 0.0 [0.0 to 100.0] | 0.0 [0.0 to 66.7]
  Treatment - Week 40: number analyzed (Participants) | 74 | 50
  Treatment - Week 40 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - Week 44: number analyzed (Participants) | 62 | 47
  Treatment - Week 44 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - Week 48: number analyzed (Participants) | 67 | 47
  Treatment - Week 48 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 52: number analyzed (Participants) | 58 | 44
  Treatment - Week 52 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 56: number analyzed (Participants) | 61 | 48
  Treatment - Week 56 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 60: number analyzed (Participants) | 47 | 39
  Treatment - Week 60 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 64: number analyzed (Participants) | 55 | 39
  Treatment - Week 64 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 68: number analyzed (Participants) | 49 | 34
  Treatment - Week 68 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 72: number analyzed (Participants) | 54 | 34
  Treatment - Week 72 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 76: number analyzed (Participants) | 42 | 29
  Treatment - Week 76 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 80: number analyzed (Participants) | 43 | 23
  Treatment - Week 80 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 84: number analyzed (Participants) | 33 | 19
  Treatment - Week 84 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 88: number analyzed (Participants) | 36 | 16
  Treatment - Week 88 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 92: number analyzed (Participants) | 30 | 13
  Treatment - Week 92 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 100.0]
  Treatment - Week 96: number analyzed (Participants) | 22 | 11
  Treatment - Week 96 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 100: number analyzed (Participants) | 18 | 10
  Treatment - Week 100 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 66.7]
  Treatment - Week 104: number analyzed (Participants) | 15 | 7
  Treatment - Week 104 | 33.33 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 108: number analyzed (Participants) | 11 | 7
  Treatment - Week 108 | 0.0 [0.0 to 66.7] | 0.0 [0.0 to 33.3]
  Treatment - Week 112: number analyzed (Participants) | 9 | 4
  Treatment - Week 112 | 0.0 [0.0 to 66.7] | 16.67 [0.0 to 33.33]
  Treatment - Week 116: number analyzed (Participants) | 4 | 2
  Treatment - Week 116 | 16.67 [0.0 to 33.33] | 16.67 [0.0 to 33.33]
  Treatment - Week 120: number analyzed (Participants) | 3 | 0
  Treatment - Week 120 | 33.33 [33.33 to 33.33] |

ADVERSE EVENTS:
Time Frame: Baseline up to 43 months
Arm/Group | Alectinib | Crizotinib
All-Cause Mortality (participants affected / at risk) | 35/152 | 40/151
Serious Adverse Events (participants affected / at risk) | 44/152 | 45/151
Other Adverse Events (participants affected / at risk) | 136/152 | 140/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=152) | Crizotinib (N=151)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Bronchopleural Fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Interstitial Lung Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 5 | 4
Lung Infection (Infections and infestations) | 3 | 0
Bronchitis (Infections and infestations) | 2 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Herpes Zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 1
Skin Infection (Infections and infestations) | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 0
Acinetobacter Infection (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Necrotising Fasciitis (Infections and infestations) | 0 | 1
Oesophageal Candidiasis (Infections and infestations) | 0 | 1
Pneumonia Klebsiella (Infections and infestations) | 0 | 1
Pyrexia (General disorders) | 1 | 3
Asthenia (General disorders) | 0 | 1
Chest Discomfort (General disorders) | 0 | 1
Hyperthermia Malignant (General disorders) | 0 | 1
Multiple Organ Dysfunction Syndrome (General disorders) | 0 | 1
Sudden Death (General disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 0
Oedema (General disorders) | 1 | 0
Aphasia (Nervous system disorders) | 0 | 1
Cerebral Haemorrhage (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 1
Epilepsy (Nervous system disorders) | 0 | 1
Hemiparesis (Nervous system disorders) | 0 | 1
Seizure (Nervous system disorders) | 0 | 1
Haemorrhage Intracranial (Nervous system disorders) | 1 | 0
Hypoglycaemic Coma (Nervous system disorders) | 1 | 0
Acute Myocardial Infarction (Cardiac disorders) | 0 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 1
Myocardial Infarction (Cardiac disorders) | 0 | 1
Sinus Bradycardia (Cardiac disorders) | 0 | 1
Cardiac Tamponade (Cardiac disorders) | 1 | 0
Pericardial Effusion (Cardiac disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 3
Vomiting (Gastrointestinal disorders) | 0 | 2
Gastrointestinal Disorder (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 0 | 1
Blood Creatinine Increased (Investigations) | 2 | 0
Alanine Aminotransferase Increased (Investigations) | 1 | 4
Aspartate Aminotransferase Increased (Investigations) | 1 | 1
Human Chorionic Gonadotropin Increased (Investigations) | 1 | 0
Deep Vein Thrombosis (Vascular disorders) | 0 | 2
Lymphoedema (Vascular disorders) | 0 | 1
Orthostatic Hypotension (Vascular disorders) | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Drug-Induced Liver Injury (Hepatobiliary disorders) | 1 | 1
Hepatic Haematoma (Hepatobiliary disorders) | 0 | 1
Hepatic Haemorrhage (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 1 | 0
Confusional State (Psychiatric disorders) | 1 | 2
Vision Blurred (Eye disorders) | 0 | 1
Forearm Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Ovarian Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal Impairment (Renal and urinary disorders) | 0 | 1
Acute Kidney Injury (Renal and urinary disorders) | 4 | 0
Urinary Retention (Renal and urinary disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Thoracic Vertebral Fracture (Injury, poisoning and procedural complications) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Uterine Polyp (Reproductive system and breast disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Oedema Peripheral (General disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alectinib (N=152) | Crizotinib (N=151)
Constipation (Gastrointestinal disorders) | 52 | 49
Nausea (Gastrointestinal disorders) | 21 | 70
Diarrohea (Gastrointestinal disorders) | 18 | 68
Vomiting (Gastrointestinal disorders) | 11 | 57
Abdominal Pain (Gastrointestinal disorders) | 9 | 7
Dyspepsia (Gastrointestinal disorders) | 5 | 12
Abdominal Pain Upper (Gastrointestinal disorders) | 8 | 6
Dysphagia (Gastrointestinal disorders) | 1 | 8
Oedema Peripheral (General disorders) | 26 | 41
Fatigue (General disorders) | 29 | 25
Asthenia (General disorders) | 11 | 11
Pyrexia (General disorders) | 7 | 9
Chest Pain (General disorders) | 9 | 5
Alanine Aminotransferase Increased (Investigations) | 22 | 42
Aspartate Aminotransferase Increased (Investigations) | 20 | 37
Blood Bilirubin Increased (Investigations) | 23 | 2
Blood Creatinine Increased (Investigations) | 11 | 6
Blood Creatine Phosphokinase Increased (Investigations) | 8 | 7
Weight Increased (Investigations) | 15 | 0
Blood Alkaline Phosphatase Increased (Investigations) | 6 | 8
Gamma-Glutamyltransferase Increased (Investigations) | 1 | 10
Dysgeusia (Nervous system disorders) | 4 | 29
Dizziness (Nervous system disorders) | 12 | 20
Headache (Nervous system disorders) | 11 | 13
Paraesthesia (Nervous system disorders) | 3 | 8
Arthralgia (Musculoskeletal and connective tissue disorders) | 17 | 10
Myalgia (Musculoskeletal and connective tissue disorders) | 24 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 12 | 7
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 6 | 10
Musculoskeletal Pain (Musculoskeletal and connective tissue disorders) | 11 | 3
Anaemia (Blood and lymphatic system disorders) | 29 | 7
Neutropenia (Blood and lymphatic system disorders) | 4 | 11
Rash (Skin and subcutaneous tissue disorders) | 16 | 14
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 11
Photosensitivity Reaction (Skin and subcutaneous tissue disorders) | 8 | 0
Visual Impairment (Eye disorders) | 2 | 18
Vision Blurred (Eye disorders) | 3 | 10
Photopsia (Eye disorders) | 0 | 9
Upper Respiratory Tract Infection (Infections and infestations) | 13 | 13
Urinary Tract Infection (Infections and infestations) | 10 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 8 | 6
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 1
Bradycardia (Cardiac disorders) | 8 | 14
Sinus Bradycardia (Cardiac disorders) | 8 | 7
Decreased Appetite (Metabolism and nutrition disorders) | 14 | 14
Insomnia (Psychiatric disorders) | 15 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02075840/Prot_001.pdf
  • Statistical Analysis Plan (2018-02-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT02075840/SAP_000.pdf